CLINICAL TRIAL: NCT04386109
Title: Neonatal Complications of Coronavirus Disease (COVID-19)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Imperial College London (Other); University of Leicester (Other); University of Nottingham (Other); University of Glasgow (Other); University Hospital of Wales (Other); Public Health England (Other Government); St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 14905
Record Dates: First submitted 2020-04-15; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-04

CONDITIONS: Neonatal COVID-19 Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neonates COVID-19 positive: 1. Neonatal COVID-19 in babies (<29 days old) in neonatal units, paediatric intensive care units and other in-patient locations.
  Interventions: Other: No intervention - exposure is to COVID-19
- Neonates born to COVID-19 positive mothers: 2. Neonates (<29 days old) born to COVID-19 positive mothers requiring neonatal care
  Interventions: Other: No intervention - exposure is to COVID-19

INTERVENTIONS:
Other: No intervention - exposure is to COVID-19 — No intervention - exposure is to COVID-19

SUMMARY:
There is an evidence gap in relation to the incidence, impact and severity of COVID-19 in newborn babies. International data are very limited, we have no robust estimates of incidence and no UK-based data with which to inform policy, clinical care, service delivery or advice to pregnant women.

The research aims are to investigate the three mains ways in which COVID-19 might affect newborns and babies that need neonatal care:

1. Newborn babies might catch COVID-19 before, during or soon after birth and this may lead to problems with breathing or feeding that need support in hospital.
2. COVID-19 could affect babies that are already on neonatal units with other medical conditions (like being very premature) that place them at greater risk of severe COVID-19.
3. COVID-19 might affect that way that pregnant women are looked after in pregnancy, labour or bith which could lead to problems for some babies, even if they do not themselves become infected with COVID-19.

DETAILED DESCRIPTION:
The investigators have established a national (UK-wide) active surveillance study using the standard British Paediatric Surveillance Unit (BPSU) approach.

Since the 1st April 2020 case notifications are being collected using the BPSU 'orange eCard' approach. Eligible babies are: neonatal COVID-19 in babies (<29 days old) in neonatal units, paediatric intensive care units and other in-patient locations and where neonates are born to COVID-19 mothers and require neonatal care. Notification cards are being sent weekly rather than the usual monthly pattern, this is so we are able to monitor case returns in 'real-time'. When paediatricians notify a case they are sent a data collection sheet which is returned complete to the BPSU-COVID-19 team at the NPEU.

The primary data collected in the study will also be cross-linking with data from: a parallel NIHR funded study of COVID-19 mothers being carried out using the UK Obstetric Surveillance System (UKOSS); MBRRACE-UK, the national surveillance of perinatal deaths; the Paediatric Intensive Care Audit Network (PICANet); and PHE England, PHS Scotland, PHS Wales and the HSC Public Health Agency Northern Ireland. This is to ensure complete case ascertainment. A later linkage will be carried out with the National Neonatal Research Database (NNRD) in order to collect more detailed clinical information.

As data are weekly reports of the findings will be generated to inform the development of policy and practice. The findings will be sent together with the UKOSS findings to: the decision makers responsible for the COVID-19 control policy at NHSE, DHSC, the Scottish, Welsh and NI governments, as well as the Royal Colleges of Paediatrics and Child Health and Obstetricians and Gynaecologists (RCPCH & RCOG respectively), and the British Association of Perinatal Medicine (BAPM). This will ensure that policy, advice to pregnant women and parents and guidance for practice benefits from the most up to date information.

Follow-up at 3 months post-notification will be carried out in order to collect the final outcomes for each baby as the first data collection will be completed when a substantial proportion of babies will still be in-patients.

Data will also be shared (subject to appropriate approvals and data sharing agreements) with the COVID-19 registries that are being developed in the UK and across Europe.

ELIGIBILITY:
Inclusion Criteria:

* Any baby:

  1. That has a diagnosis of COVID-19 made on a sample taken before 29 days of age and receives inpatient care for COVID-19 (this includes postnatal ward, neonatal unit, paediatric inpatient wards, PICU) OR
  2. Where the mother had confirmed COVID-19 at the time of birth or suspected COVID-19 at the time of birth that has subsequently been confirmed, and the baby was admitted for neonatal care

     Exclusion Criteria:

Ages: 1 Day to 29 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Babies admitted for neonatal care in: a neonatal unit, a paediatric intensive care unit or an in-patient ward.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of neonatal COVID-19 | April 2020 to March 2021
  Number of neonatal participants with COVID-19 divided by the total number of live births in the population
Incidence of vertically transmitted COVID-19 | April 2020 to March 2021
  Number of neonatal participants with COVID-19 following vertically transmission of the Coronavirus divided by the total number of live births in the population

SECONDARY OUTCOMES:
Presentation and natural history of neonatal COVID-19 | April 2020 to March 2021
  Questionnaire data
Presentation of neonates with COVID-19 positive mothers | April 2020 to March 2021
  Questionnaire data
Outcomes for neonates with COVID-19 | April 2020 to March 2021
  Proportion of neonate participants who died and the proportion who were discharged home alive.
Clinical treatment of neonatal COVID-19 | April 2020 to March 2021
  Questionnaire data
Neonatal secondary impacts of maternal COVID-19 | April 2020 to March 2021
  Questionnaire data

CONTACTS AND LOCATIONS:
Overall Officials: Professor J Kurinczuk, MBChB,MSc,MD, Principal Investigator — University of Oxford; Dr C Gale, MBBS,MSc,PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Share relevant data to international registries of neonatal COVID-19 which are being developed.
Supporting Information: Study Protocol, CSR
Time Frame: Within 6 months of the study start
Access Criteria: Funded registry with appropriate approvals to receive data